CLINICAL TRIAL: NCT02656355
Title: Gait Initiation Difficulty and Anticipatory Postural Adjustment (APA) Impairment in People With PD - Evaluation and Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103-5361B
Record Dates: First submitted 2016-01-13; First posted 2016-01-14 (Estimated); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease(PD)
Keywords: Gait Initiation; Freezing of gait; Balance training; Anticipatory postural adjustments
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Stage 1:Healthy people (No Intervention): To establish baseline and reliability.
- Stage 2:Healthy people (No Intervention): To establish stage 3 training protocol.
- Stage 2:PD people (No Intervention): To establish stage 3 training protocol.
- Stage 3:PD APA training group (Experimental): Weight shift training and APA feedback.
  Interventions: Other: Weight shift training and APA feedback
- Stage 3:PD Balance training group (Experimental): Weight shift training without APA feedback.
  Interventions: Other: Weight shift training without APA feedback
- Stage 3:PD Control group (No Intervention): Control group

INTERVENTIONS:
Other: Weight shift training and APA feedback — Use COP trajectory to train weight shift on force plate. To give APA visual feedback for subjects after weight shift training.
  Other Names: APA training group
  Arms: Stage 3:PD APA training group
Other: Weight shift training without APA feedback — Use COP trajectory to train weight shift on force plate.
  Other Names: Balance training group
  Arms: Stage 3:PD Balance training group

SUMMARY:
Gait initiation (GI) difficulty is common in people with Parkinson's disease (PD). Studies showed that the GI difficulty was related to impaired anticipatory postural adjustments (APA). In healthy people, two phases of APA related center of pressure (COP) shifting were observed before GI. In people with PD, delay and decrease amplitude of APA or abnormal multiple APAs were observed during GI.

Conventional balance tests record the maximum displacement and/or velocity of Center of pressure (COP). However, these variables could not show the performance of APA. Previous studies suggested that balance and gait initiation were controlled by separate neural circuitries. This could explain why the conventional COP measurement did not correlate to GI very well.

It is important to develop GI related APA tests and trainings. Researchers found that a perturbation applied before the COP displacement during GI could delay both GI and APA. This indicates that COP displacement has APA components. Our pilot study shows that there is a reverse direction of COP displacement before voluntary COP displacement, suggesting the existence of APA.

This three year project will evaluate the relationship of the APA of voluntary COP displacement and the APA of GI, establish the APA test for PD, and investigate the effect of APA training on GI in people with PD.

In the first year, 20 people without disability will be recruited. The APA before voluntary COP displacement test, APA before GI, and gait performance will be evaluated. In the second year, 15 people with PD and 15 healthy people will be recruited. Subjects will receive GI test, gait test, and APA before voluntary COP displacement test. The relationship between different types of APA will be established for PD and healthy people. In the third year, 30 people with PD will be randomized into APA training group, balance group, and control group. The different training effect will be evaluated especially on GI, gait performance, and freezing of gait.

This project will advance the knowledge of mechanism of GI difficulty. The result of this project can be applied to clinical rehabilitation of people with GI difficulty.

ELIGIBILITY:
Health subjects:

Exclusion Criteria:

* Musculoskeletal injuries on legs.
* Osteoporosis.

PD subjects:

Inclusion Criteria:

- Clinical diagnosis of Parkinson disease.

Exclusion Criteria:

* Musculoskeletal injuries on legs
* Osteoporosis.
* Any peripheral or central nervous system injury or disease patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Gait parameters | Baseline, 4 weeks and 8 weeks.
  Measure of changes in gait parameters by GaitRite and force plate.
Balance parameters | Baseline, 4 weeks and 8 weeks.
  Measure of changes in balance parameters by force plate.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886